CLINICAL TRIAL: NCT05316103
Title: Use of Probe-based Confocal Laser Endomicroscopy to Perform Targeted Optical Biopsy for Local Rectal Scars in Rectal Cancer Patients After Neoadjuvant Chemoradiotherapy
Brief Title: Targeted Optical Biopsy for Local Rectal Scars in Rectal Cancer Patients After Neoadjuvant Chemoradiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NFEC-2022-063
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; confocal laser endomicroscopy; optical biopsy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endoscopic biopsy and probe-based confocal laser endomicroscopy biopsy (Experimental): In this study , endoscopic biopsy and pCLE-targeted optical biopsy will be successively performed for local rectal scars in rectal cancer patients after neoadjuvant chemoradiotherapy.
  Interventions: Device: Probe-based confocal laser endomicroscopy targeted optical biopsy

INTERVENTIONS:
Device: Probe-based confocal laser endomicroscopy targeted optical biopsy — After intravenous injection of fluorescein sodium, pCLE-based targeted optical biopsy will be performed.

SUMMARY:
Currently, low concordance (36%) is found between clinical complete response and pathologic complete response in patients with rectal cancer after neoadjuvant chemoradiotherapy. Probe-based confocal laser endoscopy (pCLE) provides a promising targeted optical biopsy to evaluate the response to neoadjuvant chemoradiotherapy. The aim of this study is to investigate whether pCLE-targeted optical biopsy can improve the accuracy of preoperative endoscopic biopsy for local rectal scars in rectal cancer patients after neoadjuvant chemoradiotherapy.

DETAILED DESCRIPTION:
Patients with locally advanced rectal cancer can benefit from neoadjuvant chemoradiotherapy, and 20%-30% of patients receiving such therapy can attain a pathologic complete response, defined as the eradication of cancer cells. For those who reach pathologic complete response, a watch-and-wait strategy is supposed to be the best choice. However, low concordance (36%) was found between clinical complete response and pathologic complete response in patients with rectal cancer after neoadjuvant chemoradiotherapy. There is a compelling need to improve the consistency.

Probed-based confocal laser endoscopy (pCLE) is a novel endoscopic adjunct that allows real-time in vivo histological examination of mucosal surfaces. By using intravenous fluorescent agents, pCLE highlights certain mucosal elements that facilitate an optical biopsy in real time. It provides a promising targeted optical biopsy for local rectal scars in rectal cancer patients after neoadjuvant chemoradiotherapy.

The investigators perform this study to investigate whether pCLE-targeted optical biopsy could improve the accuracy of preoperative endoscopic biopsy for local rectal scars in rectal cancer patients after neoadjuvant chemoradiotherapy. In this study, rectal cancer patients after neoadjuvant chemoradiotherapy will be successively arranged to accept traditional endoscopic biopsy and pCLE-based targeted optical biopsy. The consistency rate will be calculated according to the postoperative pathological results.

ELIGIBILITY:
Inclusion Criteria:

1. Age from over 18 to under 80 years
2. American Society of Anesthesiology(ASA) score class I,II,or III
3. Locally advanced rectal cancer
4. Patient has completed standard neoadjuvant therapy
5. Expected surgical resection
6. Written informed consent

Exclusion Criteria:

1. Pregnant or lactating women
2. Acute renal insufficiency or stage II to IV chronic renal insufficiency
3. Patients with allergic constitution

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of pCLE-targeted optical biopsy | 7 days
  The investigators will use pCLE-targeted optical biopsy for local rectal scars in rectal cancer patients after neoadjuvant chemoradiotherapy and compare the pathological diagnosis between optical biopsy and surgically resected specimens.

SECONDARY OUTCOMES:
Sensitivity,specificity,positive predictive value and negative predictive value of pCLE targeted optical biopsy | 7 days
  The investigators will use pCLE-targeted optical biopsy for local rectal scars in rectal cancer patients after neoadjuvant chemoradiotherapy and compare the pathological diagnosis between optical biopsy and surgically resected specimens.
Complications of biopsy | 7 days
  Complications of biopsy, such as bleeding and drug allergies.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yan, M.D., Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gash KJ, Baser O, Kiran RP. Factors associated with degree of tumour response to neo-adjuvant radiotherapy in rectal cancer and subsequent corresponding outcomes. Eur J Surg Oncol. 2017 Nov;43(11):2052-2059. doi: 10.1016/j.ejso.2017.07.024. Epub 2017 Aug 10. PMID 28943178
- [Background] van der Sande ME, Maas M, Melenhorst J, Breukink SO, van Leerdam ME, Beets GL. Predictive Value of Endoscopic Features for a Complete Response After Chemoradiotherapy for Rectal Cancer. Ann Surg. 2021 Dec 1;274(6):e541-e547. doi: 10.1097/SLA.0000000000003718. PMID 31851000
- [Background] Ryan JE, Warrier SK, Lynch AC, Heriot AG. Assessing pathological complete response to neoadjuvant chemoradiotherapy in locally advanced rectal cancer: a systematic review. Colorectal Dis. 2015 Oct;17(10):849-61. doi: 10.1111/codi.13081. PMID 26260213
- [Background] Glynne-Jones R, Wallace M, Livingstone JI, Meyrick-Thomas J. Complete clinical response after preoperative chemoradiation in rectal cancer: is a "wait and see" policy justified? Dis Colon Rectum. 2008 Jan;51(1):10-9; discussion 19-20. doi: 10.1007/s10350-007-9080-8. Epub 2007 Nov 28. PMID 18043968
- [Background] Al-Mansour MR, Caycedo-Marulanda A, Davis BR, Alawashez A, Docimo S, Qureshi A, Tsuda S. SAGES TAVAC safety and efficacy analysis confocal laser endomicroscopy. Surg Endosc. 2021 May;35(5):2091-2103. doi: 10.1007/s00464-020-07607-3. Epub 2020 May 13. PMID 32405892
- [Background] Safatle-Ribeiro AV, Marques CFS, Pires C, Arraes L, Baba ER, Meirelles L, Kawaguti FS, da Costa Martins B, Lenz LT, de Lima MS, Gusmon-Oliveira CC, Ribeiro U Jr, Maluf-Filho F, Nahas SC. Diagnosis of Clinical Complete Response by Probe-Based Confocal Laser Endomicroscopy (pCLE) After Chemoradiation for Advanced Rectal Cancer. J Gastrointest Surg. 2021 Feb;25(2):357-368. doi: 10.1007/s11605-020-04878-y. Epub 2021 Jan 14. PMID 33443686